CLINICAL TRIAL: NCT04039724
Title: Clinical Trial to Compare the Pharmacokinetics and Safety/Tolerability of HCP1305 and Co-administration of HCP0605, HGP0816 in Healthy Male Volunteers
Brief Title: Pharmacokinetics of HCP1305 and Co-administration of HCP0605, HGP0816 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ALRO-102
Record Dates: First submitted 2016-02-23; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): Period 1 : HCP0605+HGP0816
  Period 2 : HCP1305
  Interventions: Drug: HCP0605 + HGP0816; Drug: HCP1305
- Sequence B (Experimental): Period 1 : HCP1305
  Period 2 : HCP0605+HGP0816
  Interventions: Drug: HCP0605 + HGP0816; Drug: HCP1305

INTERVENTIONS:
Drug: HCP0605 + HGP0816
Drug: HCP1305

SUMMARY:
To investigate the pharmacokinetics and safety/tolerability after administration of HCP1305 and co-administration of HCP0605, HGP0816 in healthy male volunteers

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetics and safety/tolerability after administration of HCP1305 and co-administration of HCP0605, HGP0816 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age 19~45 years
2. Weight is not less than 55kg, no more than 90kg and Body Mass Index(BMI) is not less than 18 kg/m2 , no more than 27 kg/m2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Subjects who judged ineligible by the investigator.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
AUClast | pre-dose(0hours), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Area under the curve to the last measurable concentration
Cmax | pre-dose(0hours), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Peak Plasma Concentration

SECONDARY OUTCOMES:
AUCinf | pre-dose(0h), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Area under the curve to infinity
Tmax | pre-dose(0hours), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Time to maximum concentration
T1/2 | pre-dose(0hours), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Terminal elimination half-life
Cl/F | pre-dose(0hours), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Apparent clearance
Vz/F | pre-dose(0hours), post-dose 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 144 hours
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea